CLINICAL TRIAL: NCT03460093
Title: Intraoperative Superior Hypogastric Plexus Block For Pain Relief During Cesarean-Section: A Prospective Case-Control Study
Brief Title: Intraoperative Superior Hypogastric Plexus Block For Pain Relief During Cesarean-Section
Status: Completed | Type: Observational
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, bahar sarıibrahim astepe, obstetrics and gynecology specialist, Kocaeli Derince Education and Research Hospital
Other Study IDs: KUGOKAEK 2017/270
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Superior Hypogastric Plexus Block
Keywords: nerve blockade; hypogastric plexus; cesarean section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case (SHPB+): Superior hypogastric plexus block present
- control (SHPB-): Superior hypogastric plexus block not present

SUMMARY:
PURPOSE: to evaluate the efficacy of superior hypogastric plexus block for pain relief after cesarean section

DETAILED DESCRIPTION:
Superior hypogastric plexus block(SHPB) for pain relief is routinely implemented in cesarean section operations at H.S.U Kocaeli Derince Education and Research Hospital. The implementation of this procedure depends on the clinical situation of the patient, the preference of the surgeon and the anesthesiologist, the course of the operation, and whether the patient wishes or not. Superior hypogastric plexus block is performed with 0.25 % bupivacaine 30 ml injected under peritoneum above promontorium.

This is a prospective case-control study. The sample consisted of 60 women having cesarean-section with general anesthesia at H.S.U Kocaeli Derince Education and Research Hospital divided into two groups: the first group having superior hypogastric plexus block for pain relief and the control group not having superior hypogastric plexus block. All participants signed an informed consent and the study was approved by the Ethics Committee of Kocaeli University ( KUGOKAEK 2017/270). The sample size was calculated with G Power 3.1 program. With ki-square Goodness-of-fit test α:0.05 ,power 95% ,effect size 0.5 total sample size was calculated 52, including 26 in case group and 26 in control group. Women having cesarean-section with spinal anesthesia, women with known bupivacaine allergy, women with anxiety-depression disorder, women with known fibromyalgia were not enrolled to the study. Age, BMI(body mass index), education status, VAS (visual analog scale) scores ,the amount of analgesic used and the hour of gas extraction and bowel movement will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women having cesarean-section operation at H.S.U Kocaeli Derince Education and Research Hospital with general anesthesia,
* Women agree to participate in the study,
* Literate women.

Exclusion Criteria:

* Women having cesarean-section with spinal anesthesia,
* Women with known bupivacaine and NSAIDS allergy,
* Women with anxiety-depression disorder,
* Women with known fibromyalgia.
* Insufficient ability to understand information in Turkish

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, pregnant, literate women having cesarean-section operation with general anesthesia at H.S.U Kocaeli Derince Education and Research Hospital Obstetrics and Gynecology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
postoperative pain score | postoperative 1. hour
  postoperative pain score evaluated with Visual Analog Scale
postoperative pain score | postoperative 6. hour
  postoperative pain score evaluated with Visual Analog Scale
postoperative pain score | postoperative 12. hour
  postoperative pain score evaluated with Visual Analog Scale
postoperative pain score | postoperative 24. hour
  postoperative pain score evaluated with Visual Analog Scale
postoperative pain score | postoperative 48. hour
  postoperative pain score evaluated with Visual Analog Scale

SECONDARY OUTCOMES:
postoperative analgesic consumption | postoperative 48 hours
  the amount of analgesic used (NSAIDs...) for pain relief after operation
postoperative passing of gas and bowel movements | postoperative 48 hours
  the hour of postoperative gas extraction and bowel movements

CONTACTS AND LOCATIONS:
Overall Officials: bahar sarıibrahim astepe, M.D, Principal Investigator — S.B.U Kocaeli Derince Education and Research Hospital
Locations (1):
- S.B.U Kocaeli Derince Education and Research Hospital, Kocaeli, Turkey (Türkiye)